CLINICAL TRIAL: NCT05185050
Title: Prevalence of Myofascial Pain Syndrome in Adolescent Idiopathic Scoliosis and the Relationship Between Myofascial Pain Syndrome and Spinal Coronal and Sagittal Alignment in Adolescent Idiopathic Scoliosis
Brief Title: Prevalence of Myofascial Pain Syndrome in Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Damla Korkmaz, Specialist Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2020.07.128
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Scoliosis; Adolescence; Myofascial Pain Syndrome; Trigger Point Pain, Myofascial; Physical Medicine and Rehabilitation
Keywords: scoliosis; sagittal alignment; cobb angle; myofascial pain
MeSH Terms: conditions — Scoliosis; Myofascial Pain Syndromes | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AIS with MPS: the participants who has Cobb angle above 10 degrees and diagnosed with myofascial pain syndrome
  Interventions: Diagnostic Test: physical examination and measurement of spinal alignment
- AIS with no pain: the participants who has Cobb angle above 10 degrees and without pain
  Interventions: Diagnostic Test: physical examination and measurement of spinal alignment

INTERVENTIONS:
Diagnostic Test: physical examination and measurement of spinal alignment — physical examination for scoliosis and myofascial pain syndrome, measurement of spinal coronal and sagittal alignment in X-ray, and pain intensity (with Visual analog scale) if necessary (for MPS group)

SUMMARY:
this is an observational and cross-sectional prevalence study. 10-18 years aged participants with adolescent idiopathic scoliosis were recruited in the study. Myofascial pain syndrome will be questioned to the participants. additionally, all participants will be evaluated using their findings for scoliosis and myofascial pain syndrome diagnostic criteria. Cobb angle, coronal balance, shoulder and pelvis asymmetry, sagittal spino-pelvic parameters of the spine (cervical lordosis, thoracic kyphosis, lumbar lordosis angles and sagittal vertical axis, sacral slop angle and pelvic incidence) will be measured.

DETAILED DESCRIPTION:
This is an observational and cross-sectional prevalence study. Patients diagnosed with adolescent idiopathic scoliosis who applied to the Physical Medicine and Rehabilitation Clinic of Kanuni Sultan Süleyman Training and Research Hospital will be included in our study. These participants will be aged between 10-18 years. These patients will be evaluated using their findings for scoliosis and myofascial pain syndrome diagnostic criteria. Cobb angle, coronal balance, shoulder and pelvis asymmetry, sagittal spino-pelvic parameters of the spine (cervical lordosis, thoracic kyphosis, lumbar lordosis angles and sagittal vertical axis, sacral slop angle and pelvic incidence) will be measured. Diagnostic criteria of Myofascial Pain Syndrome; As the Major Criteria;

1. Regional pain complaint
2. Pain or sensory change reflected from trigger points to a specific area 3. Palpable taut band in accessible muscles

4. Extreme tenderness at one point along the taut band 5. Decreased range of motion that can be measured As for the Minor Criteria;

1. Complaint of clinical pain and/or sensory change on pressurized palpation of the trigger point
2. Local twitch response of the tender point on the taut band with palpation and needling 3. Reduction of pain by injection of the tender point or stretching of the muscle Five major and at least 1 minor criteria are required for the clinical diagnosis of myofascial pain syndrome.

Patients with a previous history of surgery for scoliosis and neuromuscular scoliosis were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10-18 years
* diagnosed as adolescent idiopathic scoliosis
* agreed to participate in the study

Exclusion Criteria:

* neuromuscular or any other type of scoliosis
* any surgical treatment for scoliosis or spine.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Aged between 10-18 years with adolescent idiopathic scoliosis
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 1 day
  The Cobb angle is the most widely used measurement to quantify the magnitude of spinal deformities, especially in the case of scoliosis, on plain radiographs. Scoliosis is defined as a lateral spinal curvature with a Cobb angle of >10°
The angle of cervical lordosis | 1 day
  Cervical Lordosis refers to the natural curve of the spine in the neck, known as the cervical spine
The angle of thoracic kyphosis | 1 day
  thoracic Kyphosis is an abnormally excessive convex curvature of the spine as it occurs in the thoracic regions
The angle of lumbar lordosis | 1 day
  Lumbar lordosis is the inward curve of the lumbar, or lower, spine in the lower back
Sagittal vertical axis | 1 day
  he C7 plumb line is a radiographic reference to determine the sagittal vertical axis
pelvic incidence | 1 day
  Pelvic incidence is defined as the angle between a line perpendicular to the sacral plate at its midpoint and a line connecting this point to the femoral head axis.
sacral slope | 1 day
  Sacral slope isdefined as the angle between a sacral plate and the horizontal line. A vertical sacrum is described by a low sacral slope value and a horizontal sacrum by a high value sacral slope
pelvic tilt | 1 day
  Pelvic tilt is defined by a line through midpoint of the sacral plate and midpoint of the femoral head axes and the vertical line through the midpoint of the femoral head axis.
VAS | 1day
  Visual analog scale (The grade of pain)
Myfascial pain syndrome | 1 day
  Using by Myfascial pain syndrome diagnostic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Merve Damla Korkmaz, 1, Principal Investigator — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study Results will be shared after publication.
Time Frame: 1 day